CLINICAL TRIAL: NCT02498145
Title: Short Term Effects of Electronic Cigarettes in Tobacco Dependent Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1407014335
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-04

CONDITIONS: Smoking; Nicotine Dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine e-cigarette (Experimental): Patients will receive nicotine patch and intensive counseling plus e-cigarette with nicotine.
  Interventions: Other: Nicotine e-cigarette
- Non-nicotine e-cigarette (Active Comparator): Patients will receive nicotine patch and intensive counseling plus e-cigarette without nicotine.
  Interventions: Other: Non-nicotine e-cigarette

INTERVENTIONS:
Other: Nicotine e-cigarette — Patients will receive nicotine patch and intensive counseling plus e-cigarette with nicotine.
  Arms: Nicotine e-cigarette
Other: Non-nicotine e-cigarette — Patients will receive nicotine patch and intensive counseling plus e-cigarette without nicotine.
  Arms: Non-nicotine e-cigarette

SUMMARY:
This is a pilot human experimental study to evaluate whether the use of an e-cigarette affects lung function, exhaled CO levels, and quantitative tobacco cigarette consumption in active tobacco smokers. Subjects recruited from the Winchester Chest Clinic (WCC), Adult Primary Care Clinic (PCC) and the Smilow Cancer Hospital Smoking Cessation Service will be randomized to 1 of 2 groups: (1) nicotine patch and intensive counseling (standard care) plus nicotine e-cigarette; (2) nicotine patch and intensive counseling plus non-nicotine e-cigarette.

ELIGIBILITY:
Inclusion:

* Smoking 1 or more tobacco cigarettes per day.
* Residence within reasonable driving distance to New Haven..

Exclusion:

* Unstable psychiatric conditions such as suicidal ideation, acute psychosis, severe alcohol dependence, or dementia.
* Unstable medical conditions requiring hospitalization.
* Acute myocardial infarction or acute cerebrovascular accident within the past 30 days.
* Unstable angina.
* History of allergic reactions to adhesives.
* Women of childbearing potential who are pregnant, nursing, or not practicing effective contraception.
* Current use of an electronic cigarette.
* Subject unable or unwilling to complete study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in daily quantitative cigarette smoking | baseline, 8 weeks, and 6 months.
  Quantitative tobacco cigarette smoking will be measured by experimenter-administered rating scale for 30 days prior to treatment through 6 month follow-up.
Change in exhaled carbon monoxide (CO) levels | baseline, 8 weeks, and 6 months.
  Exhaled carbon monoxide levels will be measured with a precision instrument for detecting CO in exhaled breath.

SECONDARY OUTCOMES:
Short-term impact on lung function (spirometry) | 6 months
  Lung function will be measured by spirometry at time of study enrollment and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Baldassarri, M.D., Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States